CLINICAL TRIAL: NCT05184803
Title: A Phase 2 Study of Neoadjuvant Docetaxel, Oxaliplatin, S-1 in Patients With Unresectable Locally Advanced or Distant Metastasis Limited to Lymph Node Gastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Min-Hee Ryu, professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC2201
Record Dates: First submitted 2021-12-21; First posted 2022-01-11 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Stomach Neoplasm
Keywords: Neo-adjuvant/Adjuvant; distant metastasis limited to lymph node gastric cancer; unresectable locally advanced gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Oxaliplatin; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): treatment arm(docetaxel, oxaliplatin, S-1)
  Interventions: Drug: Docetaxel injection, oxaliplatin, S-1

INTERVENTIONS:
Drug: Docetaxel injection, oxaliplatin, S-1 — As a prior chemotherapy, intravenous administration is performed every 3 weeks for docetaxel 50 mg/m2 D1, intravenous administration for oxaliplatin 100 mg/m2 D1, and oral administration twice a day for S-140 mg/m2 D1 to 14.

SUMMARY:
Gastric cancer is the fifth most common carcinoma in the world, and cancer-related deaths rank third. It is one of the main causes of death from cancer in Korea. The cure method for gastric cancer is radical resection, but in most patients, radical resection is impossible due to local infiltration or peripheral organ or distant metastasis. Many assisted chemotherapy has been studied to improve survival rate, and in East Asia, assisted chemotherapy after complete D2 resection is the standard treatment. In the West, on the other hand, preoperative chemotherapy and postoperative assisted chemotherapy are currently standard treatments. However, due to the limited effect of adjuvant chemotherapy, it has been reported that better clinical course can be improved by increasing anticancer intensity.

In this context, a large number of prior chemotherapy have been attempted, and prior chemotherapy has several potential effects as follows. (1) Improvement of R0 resection rate due to reduced primary cancer size, (2) early treatment for micro metastasis, (3) evaluation of treatment response rate in patients with measurable lesions, and (4) unnecessary laparotomy can be avoided in patients with biologically aggressive diseases.

Based on the efficacy of chemotherapy in the combination of docetaxel, fluoropyrimidine, and platinum in metastatic gastric cancer, the investigators conducted a preceding auxiliary anti-cancer clinical trial of docetaxel, capecitabine and cisplatin in advanced gastric cancer patients who could not be completely resected by surgery. DXP was performed 4-6 cycles before surgery with the recommended dose in phase 1-2. In a total of 49 patients, R0 resection was performed in 31 (63%), and among patients, R0 resection was improved in cases where resection was not possible due to local infiltration (71%) and in cases where para-aortic node metastasis was performed (73%).

We have reported that docetaxel, oxaliplatin, and S-1 chemotherapy (DOS) as preoperative adjuvant therapy can be safely administered in combination with D2 gastrectomy and postoperative adjuvant therapy S-1 in potentially resectable local progressive gastric cancer patients. R0 resection was achieved in 97.6% of patients, and pathological complete remission was observed in 19.5%. Based on this, a phase 3 PRODIGY study was performed to evaluate the benefit of S-1 (CSC group) as a preoperative prior chemotherapy compared to S-1 (SC group) as a postoperative adjuvant therapy in gastric cancer of cT2/3N+ or cT4Nany stage, and 0.75% of the CSC group was administered HR. In the patient group undergoing surgery, the R0 resection rate was 95% in the CSC group and 84% in the SC group. In the CSC group, the pathological complete remission rate was 10.4%.

Based on these results, a clinical trial of DOS as a preoperative chemotherapy was planned for progressive gastric cancer that could not be resected due to local progression or metastasis limited to remote lymph nodes.

Primary goal: Evaluation of R0 resection rate in patients who underwent prior chemotherapy as a clinical trial.

Secondary objective: safety evaluation, overall survival period, progression-free survival period, pathological complete remission rate, and investigation of biological markers.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven metastatic gastric adenocarcinoma patients
2. As a patient who has been proven by CT to have invasion of surrounding organs (T4) according to the 8th edition of the American Joint Commission (AJCC) or confined to remote lymph nodes, the criteria for lymph node invasion are 8 mm or more in single diameter and central necrosis (rounder), (Refer to Appendix B)
3. Over 18 years old.
4. Patients with a life expectancy of at least 3 months.
5. Patients with 0 or 1 ECOG performance status
6. As defined in the relevant items below, those who have confirmed appropriate normal organ and bone marrow function:

   * Haemoglobin 9 9.0 g/dL.
   * Absolute neutrophil count (ANC) > 1.5 x 103/mCL (> 1,500 per mm3)
   * Platelet count 100 100 x 109/L
   * Serum bilirubin 1.5 1.5 x Test Laboratory Upper Limit of Normal (ULN).
   * AST(SGOT)/ALT(SGPT) 2.5 2.5x ULN of test institution.
   * Measured creatinine clearance (CL) > 40 mL/min or Cockcroft-Gault formula (Cockcroft and Gault 1976) calculated by or according to 24-hour urine samples for determining creatinine cleaning rates.

     * Male creatinine CL (mL/min) = Weight (kg)x (140-age) / 72x Serum creatinine (mg/dL)
     * Women's creatinine CL (mL/min) = Weight (kg)x (140-age) / 72 x Serum creatinine (mg/dL) x 0.85
7. A patient who has never had chemotherapy before.
8. Patients who have not previously had radiation therapy experience
9. Physical, family, social, and geographic conditions for the follow-up of patient conditions required for this study should be free of obstacles in this study.
10. Evidence of menopause or negative findings of urine or blood pregnancy response should be confirmed in premenopausal women. Women who are premenstrual for more than 12 months without any other medical cause are considered menopause. In addition, if bilateral ovarian resection, bilateral ovariectomy, and hysterectomy are performed, menopause is considered.
11. Subjects who can provide signed consent, such as compliance with the requirements and taboos specified in the test subject's consent (ICF) and this plan. Written consent must be obtained from the patient and the patient's legal representative prior to implementing the plan-related procedures, including screening evaluation.

Exclusion Criteria:

1. When pregnant women, lactating women, or pregnant women do not use appropriate contraception methods.
2. Cancer other than adenocarcinoma.
3. Patients with distant metastasis other than lymph nodes or confirmed ascites on abdominal CT before surgery.
4. History of other carcinomas or presence of pathogenic cancer (excluding non-melanoma skin cancer or cervical epithelial cancer)
5. Central nervous system metastasis.
6. Clinically significant intestinal obstruction or gastrointestinal bleeding.
7. A patient with a history of organ transplantation.
8. Active infections such as tuberculosis, hepatitis B, hepatitis C, or HIV identified by TB tests according to medical history, physical examination, radiological findings, and regional standards.

   * Tuberculosis: Tuberculosis confirmed by medical history, physical examination, or radiologically active tuberculosis, and tuberculosis tests according to regional standards (excluding active TB, old TB is acceptable)
   * Hepatitis B: If HBsAg is negative, register, and if HBsAg is positive, HBV DNA test is performed.

     * HBV DNA 500 500iu/ml (or 2500 copies/ml): Excluded
     * HBV DNA ▶500iu/ml (or 2500 copies/ml): Allow
   * Hepatitis C: If HCV Ab is negative, register, and if HCV Ab is positive, HCV RNA test is performed.

     * If HCV RNA is positive, I'll exclude it.
     * If it's HCV RNA's voice, it's allowed.
   * HIV: HIV Ag/Ab : excluding reactive faces, HIV Ag/Ab : non-reactive faces registration
9. Average QTcF (average QT interval for heart rate correction using fridericia formula) > 470 ms when calculated with three ECG tests (within 15 minutes at 2-5 minute intervals).

   If -1 test is performed and QTcF > 470 ms, 2 additional tests are performed to determine the average QTcF value.

   -If QTcF 4 470 ms after one test, no additional test is performed.
10. Other serious diseases or medical conditions.

    * Uncurable unstable heart disease, myocardial infarction within 6 months before the start of the study.
    * A history of neurological or psychiatric diseases including dementia or seizures.
    * Active, non-regulatory infection.
    * Clinically serious diarrhea.
    * Severe high calcium conditions above 12 mg/dL, which are not controlled by phonates.
    * Other serious medical conditions that may affect participation in this study.
    * Active random intravascular coagulation.
11. Patients who other researchers find inappropriate.
12. In the case of recent corticosteroids (or corresponding) treatment, except for acute hypersensitivity response therapy or low-dose (<20 mg methylprednisolone or corresponding) chronic treatment (started 6 months before the start of the study) as preventive therapy,
13. In addition to the test drug, administration of other clinical research drugs within 4 weeks or in combination.
14. Combination chemotherapy, hormone therapy, or immunotherapy.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of R0 resection rate in patients who underwent prior chemotherapy as a clinical trial. | 1 year
  Evaluation of R0 resection rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No